CLINICAL TRIAL: NCT00953173
Title: HERO Study: Helping Evaluate Reduction in Obesity
Status: Completed | Type: Observational
Sponsor: Apollo Endosurgery, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HERO Study
Record Dates: First submitted 2009-08-05; First posted 2009-08-06 (Estimated); Results first posted 2018-02-09 (Actual); Last update posted 2018-03-08 (Actual); Status verified 2018-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- LapBand: Patients who have already consented to receive the LAP-BAND AP® Adjustable Gastric Banding System
  Interventions: Device: LAP-BAND AP® Adjustable Gastric Banding System

INTERVENTIONS:
Device: LAP-BAND AP® Adjustable Gastric Banding System — The LAP-BAND AP® is a device surgically implanted via a laparoscopic procedure. It is designed to induce weight loss in severely obese patients by limiting food consumption.
  Other Names: LAP-BAND AP®

SUMMARY:
A prospective, international, multi-center study of clinical outcomes and estimated healthcare resource expenditures associated with the treatment of obesity using the LAP-BAND AP® Adjustable Gastric Banding System.

ELIGIBILITY:
Inclusion Criteria:

* Patient and investigator have made a decision, independent of the study, to proceed with LAP-BAND AP® implantation.
* Male or female aged ≥ 18 years.
* BMI ≥ 40 or a BMI ≥ 35 with one or more severe co-morbid conditions, or those who are 45.5 Kg / 100 lbs or more over their estimated ideal weight.

Exclusion Criteria:

* Prior bariatric surgery.
* Type I diabetes patients.
* Participating in another ongoing clinical study with concomitant diagnostic or therapeutic intervention that would reasonably be expected to alter patterns of care, use of medications or the outcomes under study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that have already made a decision, independent of the study, to proceed with LAP-BAND AP® implantation.
Sampling Method: Non-Probability Sample
Enrollment: 671 (Actual)
Dates: Start 2009-12; Primary Completion 2016-07 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- Everett, Washington, United States
- Adelaide, South Australia, Australia
- Jette, Belgium
- Mississauga, Ontario, Canada
- Naples, Italy
- Birmingham, United Kingdom

REFERENCES:
- [Derived] Dixon JB, Eaton LL, Curry T, Lee PC. Health Outcomes and Explant Rates After Laparoscopic Adjustable Gastric Banding: A Phase 4, Multicenter Study over 5 Years. Obesity (Silver Spring). 2018 Jan;26(1):45-52. doi: 10.1002/oby.22050. PMID 29265773
- [Derived] Lao WL, Malone DC, Armstrong EP, Voellinger D, Somers S, Jin J, Dreyer N, Globe D. Effect of adjustable gastric banding on quality of life and weight loss in the Helping Evaluate Reduction in Obesity (HERO) registry study: 2 year analysis. Curr Med Res Opin. 2015 Aug;31(8):1451-60. doi: 10.1185/03007995.2015.1059802. Epub 2015 Jul 25. PMID 26154653
- [Derived] Ponce J, Taheri S, Lusco V, Cornell C, Ng-Mak DS, Shi R, Okerson T. Efficacy and safety of the adjustable gastric band - pooled interim analysis of the APEX and HERO studies at 48 weeks. Curr Med Res Opin. 2014 May;30(5):841-8. doi: 10.1185/03007995.2013.874992. Epub 2014 Jan 16. PMID 24328415

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LapBand
Started | 671
Completed | 389
Not Completed | 282

BASELINE CHARACTERISTICS:
Arm/Group | LapBand
Number analyzed (Participants) | 652
Age, Customized [Count of Participants; unit: Participants]
  18-20 years | 9
  21-29 years | 63
  30-39 years | 164
  40-49 years | 199
  50-59 years | 166
  60+ years | 51
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 517
  Male | 135

OUTCOME MEASURES:

1. Primary Outcome: %TBWL
Description: Percent of total body weight change.
Time Frame: 5 years
Population: Patients who attended 5 year visit.
Measure: Mean (Standard Deviation); unit: % TBWL
Arm/Group | LapBand
Number analyzed (Participants) | 383
% TBWL | -18.0 (12.69)

ADVERSE EVENTS:
Time Frame: 5 Years
Arm/Group | LapBand
All-Cause Mortality (participants affected / at risk) | 2/652
Serious Adverse Events (participants affected / at risk) | 106/652
Other Adverse Events (participants affected / at risk) | 402/652
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LapBand (N=652)
Gastrointestinal Disorder (Gastrointestinal disorders) | 34 (35)
General disorders and administration site conditions (General disorders) | 2 (2)
Hepatobiliary disorder (Hepatobiliary disorders) | 1 (1)
Infections (Infections and infestations) | 3 (3)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 6 (6)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cardiac disorders (Cardiac disorders) | 9 (11)
congenital, familial and genetic disorders (Congenital, familial and genetic disorders) | 1 (2)
Eye disorders (Eye disorders) | 1 (1)
Gastrointestinal disorders-unrelated to device or procedure (Gastrointestinal disorders) | 11 (12)
General disorders-unrelated to device or procedure (General disorders) | 2 (2)
Hepatobiliary disorders-unrelated to device or procedure (Hepatobiliary disorders) | 7 (7)
infections and infestations-unrelated to device or procedure (Infections and infestations) | 8 (8)
Injury, poisoning and procedural complications-unrelated to device or procedure (Injury, poisoning and procedural complications) | 5 (5)
Metabolism and nutrition disorders-unrelated to device or procedure (Metabolism and nutrition disorders) | 3 (3)
Musculoskeletal-unrelated to device or procedure (Metabolism and nutrition disorders) | 9 (10)
Neoplasms benign, malignant and unspecified-unrelated to device or procedure (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 (12)
Nervous system-unrelated to device or procedure (Nervous system disorders) | 3 (3)
Pregnancy, puerperium and perinatal-unrelated to device or procedure (Pregnancy, puerperium and perinatal conditions) | 3 (4)
Psychiatric disorders-unrelated to device or procedure (Psychiatric disorders) | 1 (1)
Renal and urinary disorders-unrelated to device or procedure (Renal and urinary disorders) | 2 (2)
Reproductive system and breast disorders-unrelated to device or procedure (Reproductive system and breast disorders) | 2 (2)
Respiratory, thoracic and mediastinal disorders-unrelated to device or procedure (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Skin and subcutaneous tissue disorders-unrelated to device or procedure (Skin and subcutaneous tissue disorders) | 1 (1)
Surgical and medical procedures-unrelated to device or procedure (Surgical and medical procedures) | 2 (2)
Vascular disorders-unrelated to device or procedure (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LapBand (N=652)
Dysphagia (Gastrointestinal disorders) | 171 (277)
gastric polapse (Gastrointestinal disorders) | 36 (43)
Gastroesophageal reflux (Gastrointestinal disorders) | 175 (256)
Vomiting (Gastrointestinal disorders) | 205 (410)
Pouch dilatation (Injury, poisoning and procedural complications) | 41 (44)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No